CLINICAL TRIAL: NCT04366076
Title: Does a Relationship Exist Between Fetal Hiccups and Computerised Cardiotocography Parameters?
Status: Completed | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Marco La Verde, MD, research , gynecology and obstetrics, Principal Investigator, University of Campania Luigi Vanvitelli
Other Study IDs: 002
Record Dates: First submitted 2020-04-25; First posted 2020-04-28 (Actual); Last update posted 2020-05-04 (Actual); Status verified 2020-04

CONDITIONS: Fetal Conditions; Fetal Movement Disorder
Keywords: Fetal hiccups; fetal movement; computerised cardiotocography; cardiotocography; computerized analysis
MeSH Terms: interventions — Heart Rate, Fetal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- nonlaboring term singleton pregnancies: A total of 51 nonlaboring term singleton pregnancies were enrolled.
  Interventions: Diagnostic Test: Fetal heart rate (FHR) monitoring through computerized cardiotocography (cCTG) analysis antepartum

INTERVENTIONS:
Diagnostic Test: Fetal heart rate (FHR) monitoring through computerized cardiotocography (cCTG) analysis antepartum — The investigator conducted antepartum surveillance through computerized cardiotocography (cCTG) analysis antepartum. This is a non-invasive method to study fetal well being. For each patient, a cCTG was attended using a computerized cardiotocography machine. External cCTG was practised for no less than 20 min (max 60 min), two transducers were fixed on the maternal abdomen: one above the fetal heart level and the other at the uterine fundus

SUMMARY:
BACKGROUND: The physiological function of fetal hiccups and its correlation with fetal well-being is unexplored. No previous study examines the correlation between the maternal perception of the fetal hiccups and the antepartum cardiotocography.

OBJECTIVE: To evaluate the correlation between the fetal hiccups and antepartum computerised cardiotocography parameters, in nonlaboring term singleton pregnancies.

ELIGIBILITY:
Inclusion Criteria:

* physiological nonlaboring term singleton pregnancies

Exclusion Criteria:

* . Gestations complicated by fetal malformations, stillbirth, preterm deliveries or patients with missing data were excluded.

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: physiological nonlaboring term singleton pregnancies (>37 weeks) without maternal or fetal complication
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-04-20 (Actual); Study Completion 2020-04-20 (Actual)

PRIMARY OUTCOMES:
The primary outcome was the correlation between the fetal hiccups and antepartum computerised cardiotocography parameters, in nonlaboring term singleton pregnancies. | pre-intervention
  antepartum computerised cardiotocography parameters are the baseline fetal heart rate (Basal FHR), accelerations and decelerations, long-term FHR variation (LTV), short-term FHR variation (STV), episodes of high/low FHR variation and number of fetal movements for an hour (FM)

CONTACTS AND LOCATIONS:
Locations (1):
- Università degli studi della Campania "Luigi Vanvitelli"- OB & Gyn -, Napoli, Italia, Italy

IPD SHARING:
Plan to Share IPD: Undecided